CLINICAL TRIAL: NCT01961908
Title: A Phase 2, Multi-Center, Open-Label Extension Study to Evaluate the Safety and Efficacy of 12 mg Proellex® (Telapristone Acetate) Administered Orally in the Treatment of Premenopausal Women With Confirmed Symptomatic Endometriosis
Brief Title: Open-Label Extension Study to ZPE-202
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZPE-202EXT
Record Dates: First submitted 2013-10-10; First posted 2013-10-14 (Estimated); Last update posted 2014-02-07 (Estimated); Status verified 2014-02

CONDITIONS: Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — telapristone acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 12 mg Proellex (Experimental): 12 mg capsules, orally, once daily for 8 months, including off-drug interval
  Interventions: Drug: Proellex

INTERVENTIONS:
Drug: Proellex
  Other Names: telepristone acetate

SUMMARY:
This study is a phase 2, open-label extension study of 12 mg Proellex for 2 treatment cycles, each with a 16 week active dosing period. Endometriosis pain, dysmenorrhea, non-menstrual pelvic pain and dyspareunia (BBSS) as well as use of pain medications, and vaginal bleeding intensity will be recorded using an electronic diary and Visual Analog Scale (VAS) pain assessment will be utilized. All subjects will have completed an Off-Drug Interval (ODI) prior to starting treatment. Visit 1 will be scheduled within a week before the next expected menses (+/- 2 days), following the off-drug interval. Subjects will receive 2 cycles of treatment separated by an off-drug interval (ODI), after which they will be followed until menses has returned. During the follow-up period subjects will continue to record study information in the electronic diary. The final follow-up visit will be scheduled after blood flow has stopped.

ELIGIBILITY:
Inclusion Criteria:

* Successful completion of protocol ZPE-202, or subject who withdrew from ZPE-202 for lack of efficacy after completion of at least 28 days of double-blind treatment (after Visit 3)
* Agreement not to attempt to become pregnant during the trial
* Women of child-bearing potential must be willing to use double-barrier contraception during the study and for 30 days after discontinuation of study medication. Acceptable double-barrier methods are: male condom with spermicide; male condom with diaphragm; diaphragm containing spermicide plus additional intra-vaginal spermicide
* Has a negative pregnancy test at Visit 1
* Is available for all treatment and follow-up visits

Exclusion Criteria:

* Subject is pregnant or lactating or is attempting or expecting to become pregnant during the 6-7 month study period
* Concurrent use of any testosterone, progestin, androgen, estrogen, anabolic steroids, dehydroepiandrosterone (DHEA) or hormonal products for at least 2 weeks prior to Visit 1.
* Presence of intramural fibroids that impact the endometrial stripe, submucosal fibroids (any size), or endometrial polyps. Subserosal and intramural fibroids with no impact on the endometrial stripe are acceptable.
* Presence of endometrioma(s)
* Present history or condition that causes non-endometriosis related dyspareunia (e.g. vulvar vestibulitis).
* Past or present history of thrombophlebitis or thromboembolic disorders.
* Known or suspected carcinoma of the breast or reproductive organs.
* Cervical dysplasia classified as Atypical Squamous Cells of Undetermined Significance (ASCUS) associated with high-risk human papilloma virus (HPV) or Low/High Grade Squamous Intraepithelial Lesion (LGSIL or HGSIL).
* Known active infection with HIV, Hepatitis A, B or C.
* Endometrial stripe ≥18 mm in thickness at Visit 1.
* Subject is currently taking cimetidine or spironolactone.
* Clinically significant abnormal findings on screening examination and laboratory assessments or any condition which in the opinion of the investigator would interfere with the participant's ability to comply with the study instructions or endanger the participant if she took part in the study.

Ages: 18 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2013-12; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
Prescription Analgesic Use | 10 months
  Percent change from baseline in use of prescription analgesics comparing the ZPE-202 baseline nominal 28-day menstrual cycle (including menstrual event) to a similar period leading up to the end of treatment in the extension study (Visit 10)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Little Rock, Arkansas
  - Clearwater, Florida
  - Margate, Florida
  - Summerville, South Carolina
  - Houston, Texas
  - Riverton, Utah
  - Salt Lake City, Utah

REFERENCES:
- See also: Sponsor Corporate Website — http://www.reprosrx.com